CLINICAL TRIAL: NCT06395922
Title: Blockbuster LMA Versus Baska Mask in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Clinical Trial
Brief Title: Blockbuster LMA Versus Baska Mask in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rabab Mohamed Mohamed Mohamed, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 36264PR526/2/24
Record Dates: First submitted 2024-04-27; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Blockbuster LMA; Baska Mask; Laparoscopic Cholecystectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blockbuster LMA (Group BL) (Experimental): The LMA was inserted using the recommended technique, with the patient's head in the sniffing position. The appropriate size was selected based on body weight (size 3 for 30-50 kg, size 4 for 50-70 kg).
  Interventions: Device: Blockbuster LMA
- Baska Mask (Group BM) (Experimental): The BM was inserted by opening the mouth, avoiding the tongue, and negotiating the palatopharyngeal curve using the hand-tab.
  Interventions: Device: Baska Mask

INTERVENTIONS:
Device: Blockbuster LMA — The LMA was inserted using the recommended technique, with the patient's head in the sniffing position. The appropriate size was selected based on body weight (size 3 for 30-50 kg, size 4 for 50-70 kg)
  Arms: Blockbuster LMA (Group BL)
Device: Baska Mask — The BM was inserted by opening the mouth, avoiding the tongue, and negotiating the palatopharyngeal curve using the hand-tab.
  Arms: Baska Mask (Group BM)

SUMMARY:
This study aimed to compare the performance and safety profiles of two supraglottic airway devices (SADs), the Blockbuster laryngeal mask airway (LMA) and the Baska Mask (BM), in patients underwent laparoscopic cholecystectomy (LC).

DETAILED DESCRIPTION:
Laparoscopic surgery has become increasingly prevalent across numerous surgical disciplines due to the well-established benefits it offers over traditional open procedures. Laparoscopic cholecystectomy (LC), the surgical removal of the gallbladder, stands out as one of the most frequently performed laparoscopic operations worldwide.

Supraglottic airway devices (SADs) play a crucial role in airway management algorithms, serving as viable alternatives in both anticipated and unanticipated difficult airway situations.

The laryngeal mask airway (LMA) can be utilized to establish a routine airway during general anesthesia or, less frequently, as a conduit for tracheal intubation. Newer, improved LMA designs incorporate cuffs that provide higher sealing pressures than classic LMAs, while also allowing for the venting of gastric contents through a dedicated drain tube.

The Baska Mask (BM), a second-generation SAD, features a non-inflatable cuff that is continuous with the airway channel, thereby inflating with positive pressure ventilation to improve cuff seal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Scheduled for elective LC under general anesthesia.

Exclusion Criteria:

* Anticipated difficult airway.
* Renal dysfunction.
* Hiatus hernia.
* Obesity.
* Pregnancy.
* Patients taking rate-controlling medications, steroids, opioids, or regular antacids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 30 min after insertion
  Oropharyngeal leak pressure was measured Just after insertion and 30 min after insertion.

SECONDARY OUTCOMES:
Device insertion time | 5 min after insertion
  The time from start of insertion till successful insertion.
The incidence of successful gastric tube placement | 10 min after insertion
  The incidence of successful gastric tube placement through the device.
Complications | 24 hours postoperatively
  Complications such as including pain in the throat, difficulty in swallowing, cough, and blood on the device were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.